CLINICAL TRIAL: NCT05059223
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi- Center Study to Assess the Efficacy and Safety of AXS-12 in the Treatment of Cataplexy and Excessive Daytime Sleepiness in Subjects With Narcolepsy
Brief Title: A Study to Assess the Efficacy and Safety of AXS-12 (Reboxetine) in Patients With Narcolepsy
Acronym: SYMPHONY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-12-301
Record Dates: First submitted 2021-09-09; First posted 2021-09-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Narcolepsy; Cataplexy; Excessive Daytime Sleepiness
Keywords: AXS-12; Narcolepsy; Cataplexy; Excessive daytime sleepiness; Reboxetine; Axsome
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence | interventions — Reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-12 (reboxetine) (Experimental): Up to 5 weeks
  Interventions: Drug: AXS-12 (reboxetine)
- Placebo (Placebo Comparator): Up to 5 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-12 (reboxetine) — AXS-12 tablets, taken twice daily
  Arms: AXS-12 (reboxetine)
Drug: Placebo — Placebo tablets, taken twice daily
  Arms: Placebo

SUMMARY:
This study is a multi-center, double-blind, placebo-controlled, randomized Phase 3 trial to assess the safety and efficacy of AXS-12 in narcoleptic subjects with cataplexy and excessive daytime sleepiness (EDS).

DETAILED DESCRIPTION:
Eligible subjects must have a diagnosis of narcolepsy per the International Classification of Sleep Disorders (ICSD-3), and exhibit symptoms of both cataplexy and EDS. Subjects meeting the entry criteria will be randomized in a 1:1 ratio to receive either AXS-12 or placebo for five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 15 and 75 years of age, inclusive
* Primary diagnosis of narcolepsy with cataplexy
* Willing and able to comply with the study requirements

Exclusion Criteria:

* Other clinically significant conditions potentially causing EDS
* Clinically significant psychiatric disorders

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Frequency of cataplexy attacks | Change from Baseline to Week 5
  Average number of cataplexy attacks per week

CONTACTS AND LOCATIONS:
Locations (48):
- United States (46):
  - Clinical Research Site, Alabaster, Alabama
  - Clinical Research Site, Peoria, Arizona
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Redwood City, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Santa Monica, California
  - Clinical Research Site, Boulder, Colorado
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Clearwater, Florida
  - Clinical Research Site, Doral, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, St. Petersburg, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Winter Park, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Gainesville, Georgia
  - Clinical Research Site, Macon, Georgia
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Honolulu, Hawaii
  - Clinical Research Site, Peoria, Illinois
  - Clinical Research Site, Fort Wayne, Indiana
  - Clinical Research Site, Chevy Chase, Maryland
  - Clinical Research Site, Newton, Massachusetts
  - Clinical Research Site, North Dartmouth, Massachusetts
  - Clinical Research Site, Kalamazoo, Michigan
  - Clinical Research Site, Novi, Michigan
  - Clinical Research Site, Maplewood, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, West Long Branch, New Jersey
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, New Hyde Park, New York
  - Clinical Research Site, Denver, North Carolina
  - Clinical Research Site, Gastonia, North Carolina
  - Clinical Research Site, Huntersville, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Wyomissing, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Columbia, South Carolina
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Sugar Land, Texas
  - Clinical Research Site, Williamsburg, Virginia
- Canada (2):
  - Clinical Research Site, Markham, Ontario
  - Clinical Research Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SYMPHONY Study Website — http://SYMPHONYstudy.com
- See also: Axsome Therapeutics Website — http://www.axsome.com